CLINICAL TRIAL: NCT06643221
Title: Exercise-induced Adrenergic Receptor Signaling as an Immune Adjuvant for Allogeneic Cell Therapies
Brief Title: Exercise as an Immune Adjuvant for Allogeneic Cell Therapies
Acronym: Allo-X
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1801161041; 5R01CA277493-02 (NIH)
Record Dates: First submitted 2024-10-08; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Leukemia; Hematopoetic Stem Cell Transplantation; Donor Lymphocyte Infusion; CAR T-Cell Therapy; Lymphoma; Cell Therapy
Keywords: exercise; cell therapy; beta-blockers; immune function; phosphodiesterase inhibitor; CAR T-cells; NK-cells; cytokine-induced killer cells; cytokine-induced memory-like NK-cells; monoclonal antibodies; leukemia; lymphoma; donor lymphocyte infusion; gamma-delta T-cells
MeSH Terms: conditions — Leukemia; Lymphoma; Motor Activity | interventions — Exercise; Isoproterenol; Bisoprolol; Nadolol; Carvedilol; Roflumilast; Tablets

STUDY DESIGN:
Intervention Model Description: This trial has two main approaches:
  1. Single Group - Blood samples collected from healthy participants during and after an acute exercise bout (or isoproterenol infusion) are compared to the 'resting' sample of the donor.
  2. Crossover - Blood samples collected from healthy participants during and after an acute bout of exercise (or isoproterenol infusion) are compared across different conditions involving a placebo, selective beta-antagonists, non-selective beta-antagonists and phosphodiesterase inhibitors. In this model, all participants act as their own controls and a wash out period of at least 7-days is interspersed between each trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Exercise Cohort (Experimental): After an initial maximal graded exercise test to determine maximal oxygen uptake and peak cycling power, healthy participants will undergo a 20-minute graded exercise test at intensities corresponding to 50, 60, 70 and 80% VO2max (5-minutes per stage)
  Interventions: Behavioral: Exercise
- Exercise + Beta Blocker Cohort (Placebo Comparator): Healthy participants will complete a 20-minute graded exercise test at intensities ranging from 50-80-% of the maximal oxygen uptake under the following conditions: (1) Placebo; (2) 10mg bisoprolol ingestion; (3) 80ng nadolol ingestion; (4) 50ng carvedilol ingestion; (5) 10mg bisoprolol + 100mcg roflumilast ingestion. All drugs and placebo will be ingested 2-3h prior to exercise. Trial conditions will be double-blind and cross over with each participant serving as their own cntrol
  Interventions: Drug: Placebo; Drug: Bisoprolol Fumarate Tablet 10 mg; Drug: Nadolol (1 x 80 mg) Tablets (Invamed, Inc); Drug: Carvedilol 50 mg; Drug: Roflumilast 500 Mcg Oral Tablet
- Isoproterenol Infusion Cohort (Experimental): To determine if pharmacological activation of beta-adrenergic receptors evokes an immune respponse akin to exercise, healthy participants will receive an intravenous infusion of isoproterenol (50ng/kg/min)
  Interventions: Drug: Isoproterenol

INTERVENTIONS:
Behavioral: Exercise — After an initial maximal graded exercise test to determine maximal oxygen uptake and peak cycling power, healthy participants will undergo a 20-minute graded exercise test at intensities corresponding to 50, 60, 70 and 80% VO2max (5-minutes per stage)
  Arms: Exercise Cohort
Drug: Isoproterenol — To determine if pharmacological activation of beta-adrenergic receptors evokes an immune respponse akin to exercise, healthy participants will receive an intravenous infusion of isoproterenol (50ng/kg/min)
  Arms: Isoproterenol Infusion Cohort
Drug: Placebo — Healthy participants will consume the placebo 2-3h prior to completing a 20-minute graded exercise test at intensities ranging from 50-80-% of the maximal oxygen uptake
  Arms: Exercise + Beta Blocker Cohort
Drug: Bisoprolol Fumarate Tablet 10 mg — Healthy participants will consume a 10mg Bisoprolol Fumerate tablet 2-3h prior to completing a 20-minute graded exercise test at intensities ranging from 50-80-% of the maximal oxygen uptake
  Arms: Exercise + Beta Blocker Cohort
Drug: Nadolol (1 x 80 mg) Tablets (Invamed, Inc) — Healthy participants will consume a 80mg Nadolol tablet 2-3h prior to completing a 20-minute graded exercise test at intensities ranging from 50-80-% of the maximal oxygen uptake
  Arms: Exercise + Beta Blocker Cohort
Drug: Carvedilol 50 mg — Healthy participants will consume a 50mg Carvedilol tablet 2-3h prior to completing a 20-minute graded exercise test at intensities ranging from 50-80-% of the maximal oxygen uptake
  Arms: Exercise + Beta Blocker Cohort
Drug: Roflumilast 500 Mcg Oral Tablet — Healthy participants will consume a 500mcg Roflumilast tablet and a 10mg Bisoprolol tablet 2-3h prior to completing a 20-minute graded exercise test at intensities ranging from 50-80-% of the maximal oxygen uptake
  Arms: Exercise + Beta Blocker Cohort

SUMMARY:
This study aims to improve the treatment of blood cancer by using exercise to collect healthier immune cells from donors. Allogeneic adoptive cell therapy is a treatment where immune cells from a healthy donor are given to a cancer patient, usually to help prevent or treat cancer relapse after a stem cell transplant. These donor cells can either be directly infused into the patient or grown in a lab to create more specialized immune cells that target and kill cancer. While this therapy has been helpful for many patients, there is a need to make it more effective for a larger group and reduce side effects like graft-versus-host disease (GvHD), where the donor's immune cells attack the patient's healthy tissue.

This Early Phase 1 trial will test whether exercise can help produce better immune cells from donors. The investigators will recruit healthy participants for three study groups:

1. Exercise Group: Participants will complete a 20-minute cycling exercise session. The investigators will collect blood samples before, during, and after exercise to study the number and quality of immune cells. The investigators will also use the collected cells to create immune therapies and test their ability to kill cancer cells in the lab and control cancer growth in mice.
2. Exercise and Beta Blocker Group: In this group, participants will complete up to five cycling sessions, with at least a week between each session. Before each session, participants will take either a placebo or a drug (beta blocker) that blocks stress hormones like adrenaline. The investigators will collect blood samples before and during exercise to see how blocking these hormones changes the effect of exercise on immune cells.
3. Isoproterenol Group: Participants in this group will receive a 20-minute infusion of isoproterenol, a drug that mimics the effects of adrenaline. The investigators will collect blood samples before, during, and after the infusion to see if the drug causes similar immune changes to those caused by exercise.

Participants can join one, two, or all three groups. This research will help understand whether exercise can improve immune cell therapies for treating blood cancer and reduce the risk of GvHD, making these treatments safer and more effective.

DETAILED DESCRIPTION:
Background:

Allogeneic cell therapies encompass various approaches, including donor lymphocyte infusions (DLI) and engineered immune cell products like chimeric antigen receptor (CAR) T-cells, gamma delta (γδ) T-cells, cytokine-induced killer (CIK) cells, and cytokine-induced memory-like natural killer (NK) cells. These therapies are commonly employed after allogeneic hematopoietic cell transplantation (alloHCT) to prevent or treat leukemic relapse in high-risk patients. However, while these therapies have shown potential, the success rates for DLI and expanded cell products remain limited. DLI, in particular, carries the risk of inducing graft-versus-host disease (GvHD), where donor T-cells attack healthy tissues, leading to significant morbidity. Furthermore, expanded cell products face challenges related to manufacturing times, efficacy, and cost, which can limit their accessibility and effectiveness. Therefore, there is a critical need to enhance the graft-versus-leukemia/lymphoma (GvL) effects of DLI and improve the efficacy of expanded cell products to achieve better outcomes for a larger number of patients without increasing the risk of GvHD, thereby broadening their use in clinical practice.

Exercise has been shown to contribute to lower cancer risk, improve outcomes in cancer survivors, and act as an adjuvant for several cancer therapies. The present exercise model involves an acute single bout of moderate to vigorous intensity exercise lasting 20 minutes, which evokes a catecholamine-dependent mobilization and redistribution of effector lymphocytes (e.g., natural killer cells, γδ T-cells, and CD8+ T-cells). This response may enhance long-term immunosurveillance by improving the recognition and destruction of premalignant cells and contributing to the suppression of tumor growth. The overarching research question is: Can lymphocytes be collected from blood during the exercise-induced mobilization phase to generate superior cell products for cancer immunotherapy? The overall vision is to develop exercise-mobilized lymphocytes into a therapy that increases the efficacy of both DLI and expanded cell products (e.g., CAR T-cells, γδ T-cells, CIK cells, and cytokine-induced memory-like NK cells) for treating leukemia/lymphoma relapse. This novel approach, termed "DLI-X," has the potential to improve a pre-existing therapy for the treatment of blood cancers at minimal cost.

The goals of this proposal are to conduct head-to-head comparisons between standard DLI and DLI-X, both in vitro and in xenogeneic mouse models engrafted with various human hematological cancers, and to identify the underlying mechanisms driving the enhanced anti-leukemia/lymphoma response of DLI-X.

The overarching hypothesis is that DLI-X and the expanded cell products manufactured from these exercise-mobilized lymphocytes will exhibit enhanced GvL effects against multiple hematological malignancies compared to standard DLI. These effects will be driven by β2-adrenergic receptor (β2-AR)-mediated transcriptomic and proteomic changes that promote target cell recognition and cytotoxicity. Additionally, it is proposed that DLI-X will improve the efficacy of combination therapies such as blinatumomab, a bi-specific T-cell engager, and monoclonal antibodies designed to increase antibody-dependent cellular cytotoxicity (ADCC), thereby enhancing tumor growth suppression and the GvL effects of DLI.

Specific Aims:

1. Evaluate how acute, single bouts of moderate to vigorous intensity exercise lasting 20 minutes influence the number, phenotype, and molecular characteristics of immune cells in the blood.
2. Determine whether immune cells collected post-exercise yield superior therapeutic products compared to those collected under resting conditions from the same donor.
3. Investigate the role of adrenergic receptor signaling in mediating these effects

Procedures:

Healthy participants will be recruited into three distinct arms (cohorts) of this study: (1) Exercise Cohort; (2) Exercise + Beta Blocker Cohort; and/or (3) Isoproterenol Infusion Cohort. Participants may enroll in one, two, or all three study arms. The procedures for each cohort are outlined below.

Exercise Cohort Participants in the Exercise Cohort will be scheduled to visit the laboratory for three separate sessions between 08:00 and 10:00. During each visit, staff will confirm adherence to pre-testing guidelines (e.g., 8-12 hours of fasting and no vigorous physical activity). Any participant who does not meet these guidelines will be rescheduled.

Exercise Cohort Visit 1: Screening and Graded Exercise Test Time Commitment: 60 minutes

1. Informed Consent: A member of the research team will obtain written informed consent from the participant.
2. Pre-screening Questionnaire: Participants will complete the AHA/ACSM pre-screening questionnaire to verify that inclusion and exclusion criteria are met.
3. Anthropometric Measurements: Height and weight will be measured.
4. Blood Samples: A fingerstick capillary blood sample will be collected (using a sterile spring-loaded lancet) for total cholesterol and fasting glucose quantification, using an automated handheld analyzer (Cardiocheck).
5. Blood Pressure Measurement: Resting blood pressure will be measured using a manual or automated blood pressure cuff.
6. Risk Stratification: Participants deemed ineligible after screening will be excluded from further participation.
7. Graded Exercise Test: Participants will perform a maximal exercise protocol on an indoor stationary bicycle. They will wear a heart rate monitor and a face mask connected to a metabolic cart for continuous measurement of heart rate and respiratory gases. The test will begin at 50 Watts for females and 75 Watts for males, with power increased by 15 Watts each minute until exhaustion. Maximal oxygen uptake (VO2max), ventilatory threshold, and peak cycling power will be determined.

Exercise Cohort Visits 2 and 3 Time Commitment: 2 hours per visit Participants will return to the laboratory 3-10 days after Visit 1 and 7-14 days after Visit 2.

1. Pre-Exercise Procedures: An IV catheter will be inserted into a peripheral arm vein by a trained phlebotomist. A pre-exercise blood sample (approximately 120 mL) will be collected.
2. Exercise Protocol: Participants will engage in a 20-minute session of moderate-to-vigorous cycling exercise at power outputs corresponding to 50%, 60%, 70%, and 80% of their predetermined maximal oxygen uptake (VO2max) for 5-minute increments. Participants will not be exercised to exhaustion during these trials. Blood pressure measurements and ratings of perceived exertion will be collected every 5 minutes during the exercise session and immediately after.
3. Blood Sampling During Exercise: Additional venous blood samples (total volume during exercise: 80 mL) will be collected through the IV catheter at various stages of the exercise protocol.
4. Post-Exercise Blood Draw: A final blood draw of 15 mL will be collected 1 hour post-exercise.

Total Blood Volume: Participants will donate a total of 215 mL of blood (120 mL pre-exercise, 80 mL during exercise, and 15 mL post-exercise) per visit, for a total of 430ml across both visits. Additionally, several droplets of capillary blood (approximately 10-20 µL) will be collected during Visit 1 for screening purposes.

The procedures for Visits 2 and 3 will be identical. The rationale for two visits is to obtain sufficient blood to generate multiple therapeutic cell products from the same donor. The total time commitment for this cohort is approximately 5 hours.

Exercise + Beta Blocker Cohort

Time Commitment: 21 hours Participants in the Exercise + Beta Blocker Cohort will be scheduled to visit the laboratory for six separate sessions between 08:00 and 10:00, which will be spread over 6-10 weeks. During each visit, study staff will confirm adherence to pre-testing guidelines (e.g., 8-12 hours of fasting and no vigorous physical activity). Any participant who does not meet these guidelines will be rescheduled.

Exercise + Beta Blocker Cohort Visit 1 - Graded Exercise Test Time Commitment: 60 minutes. Participants will complete a graded exercise test on an indoor stationary bicycle to determine their maximal oxygen uptake (VO₂max) and peak cycling power. This test will ensure the appropriate intensity levels for subsequent exercise trials.

Exercise + Beta Blocker Cohort Visits 2-6 - Exercise Trials Time Commitment: 20 hours

The remaining five visits will consist of the main exercise trials, where participants will undergo the following procedures. There will be a 7-10 day period between each exercise trial visit to allow for recovery and minimize potential carryover effects from the drugs administered:

1. Drug Administration: The drug trials will be conducted in a block, randomized double-blind setting to ensure that neither the experimenter nor the participant knows which trial is occurring. The randomization will be computed by a member of the research team not involved in performing the exercise trials. The timing of drug administration is based on peak plasma concentrations of each drug. At 3 hours, 2 hours, and 1 hour prior to each exercise trial, participants will be administered either a drug or a placebo pill according to the following outline:

   Trial 1: Placebo at all time points Trial 2: Nadolol at 3 hours Placebo at 2 hours and 1 hour Trial 3: Bisoprolol at 3 hours Placebo at 2 hours and 1 hour Trial 4: Placebo at 3 hours and 1 hour, Carvedilol at 2 hours Trial 5: Bisoprolol at 3 hours, Placebo at 2 hours, Roflumilast at 1 hour
2. Pre-Drug Procedures: Prior to the ingestion of the drug or placebo, an IV catheter will be inserted into a peripheral arm vein by a trained phlebotomist. A pre-drug blood sample will be collected.
3. Post-Drug, Pre-Exercise Blood Sample: After the drug or placebo has been ingested and 30 minutes before exercise begins, a post-drug, pre-exercise blood sample will be collected.
4. Exercise Protocol: Participants will engage in a 20-minute session of moderate-to-vigorous cycling exercise at power outputs corresponding to 50%, 60%, 70%, and 80% of their predetermined VO₂max for 5-minute increments. Participants will not be exercised to exhaustion during these trials. Blood pressure measurements and ratings of perceived exertion will be collected every 5 minutes during the exercise session and immediately after.
5. Blood Sampling During Exercise: Additional venous blood samples will be collected through the IV catheter at various time points throughout the exercise protocol.
6. Post-Exercise Recovery Blood Samples: Additional blood samples will be collected during the recovery phase, at various time points ranging from 5 to 60 minutes post-exercise.

Total Blood Volume: Participants in this cohort will donate a total of approximately 220 mL of blood per visit. The cumulative total blood volume for this cohort across all six visits is approximately 1,320 mL.

Isoproterenol Cohort Participants in the Isoproterenol Cohort will be scheduled to visit the laboratory for three separate sessions between 08:00 and 10:00. During each visit, study staff will confirm adherence to pre-testing guidelines (e.g., 8-12 hours of fasting and no vigorous physical activity). Any participant who does not meet these guidelines will be rescheduled.

Isoproterenol Cohort Visit 1: Screening and Isoproterenol Infusion Time Commitment: 2 hours

1. Informed Consent: A member of the research team will obtain written informed consent from the participant.
2. Pre-screening Questionnaire: Participants will complete the AHA/ACSM pre-screening questionnaire to verify that inclusion and exclusion criteria are met.
3. Anthropometric Measurements: Height and weight will be measured.
4. Blood Samples: A fingerstick capillary blood sample will be collected (using a sterile spring-loaded lancet) for total cholesterol and fasting glucose quantification, using an automated handheld analyzer (Cardiocheck).
5. Blood Pressure Measurement: Resting blood pressure will be measured using a manual or automated blood pressure cuff.
6. Risk Stratification: Participants deemed ineligible after screening will be excluded from further participation.
7. Pre-Infusion Procedures: The participant will be fitted with electrodes attached to an electrocardiogram (ECG; 12-lead) and will receive a resting ECG reading, which will be monitored by a physician cardiologist. The cardiologist will make the decision whether to proceed with the infusion or exclude the participant from the study. Two IV catheters will be inserted into bilateral peripheral arm veins by a trained phlebotomist. One catheter will be used for delivering isoproterenol, and one will be used for collecting blood samples. A pre-infusion blood sample (approximately 120 mL) will be collected.
8. Isoproterenol Infusion Protocol: Participants will receive a continuous infusion of isoproterenol for 20-minutes at a concentration of 50ng/min/kg. Blood pressure measurements will be collected every 5 minutes during the infusion and ECG activity will be monitored continuously. A physician cardiologist will monitor the entire infusion procedure.
9. Blood Sampling During Infusion: Additional venous blood samples (total volume during exercise: 80 mL) will be collected through the IV catheter during the last 5-minutes of the infusion protocol.
10. Post-Infusion Blood Draw: A final blood draw of 15 mL will be collected 1 hour post-exercise.

Total Blood Volume: Participants will donate a total of 215 mL of blood (120 mL pre-infusion, 80 mL during infusion, and 15 mL post-infusion) during this visit. Additionally, several droplets of capillary blood (approximately 10-20 µL) will be collected during Visit 1 for screening purposes.

Outcome Measures:

The outcome measures for all three cohorts will be identical as described in the 'Outcome Measures' section of this protocol

ELIGIBILITY:
Procedures are in place for protecting against or minimizing the risks to the healthy volunteers recruited for this study. Physical risk to volunteers and matched related donors will be protected through health screening to determine study eligibility, and medical monitoring with an established test termination criterion during the exercise and isoproterenol infusion trials.

To protect against the remote risk of an adverse cardiac event occurring during exercise and isoproterenol infusion, the study will only enroll volunteers who are considered "low risk" for maximal stress testing in accordance with the guidelines published by the American College of Sports Medicine (ACSM) and American Heart Association (AHA). Individuals who are considered "low risk" are men and women who are asymptomatic and have no more than one risk factor for cardiovascular disease (CVD). The risks to subjects are therefore extremely low. All infusions will take place in the Clinical and Translational Sciences Research Center (CATS) Infusion Suite, which is a designated University of Arizona campus facility for infusion trials and equipped with appropriate medical personnel and monitoring equipment (i.e. ECG). The graded exercise tests and isoproterenol infusions procedures will be performed under the direction of a licensed and board-certified cardiologist

Inclusion Criteria:

Participants must:

* Be between 21 and 55 years of age.
* Be classified as 'low-risk' for graded exercise/stress testing according to ACSM-AHA criteria.
* Have no contraindications for the use of isoproterenol, carvedilol, bisoprolol, nadolol, or roflumilast as per FDA guidelines.

Exclusion Criteria:

Participants will be excluded if they:

* Currently use tobacco products or have quit within the last 6 months.
* Have a body mass index (BMI) greater than 34 kg/m² or waist circumference exceeding 102 cm for men and 88 cm for women.
* Use any medications known to affect the immune system or regularly take ibuprofen/aspirin, antidepressants, or medications that alter blood pressure or cardiovascular function.
* Use of hormone replacement therapy.
* Are pregnant or breastfeeding.
* Have chronic or debilitating arthritis or have been bedridden in the past three months.
* Experienced a common illness (e.g., colds) within the past 6 weeks.
* Have central or peripheral nervous disorders, a history of stroke, or major affective disorder.
* Are infected with HIV or hepatitis or have any autoimmune disease.
* Have known cardiovascular disease or contraindications for the use of isoproterenol, carvedilol, bisoprolol, nadolol, or roflumilast.
* Use any prescription medications or have an allergy to beta-blockers.
* Have a resting heart rate of less than 50 beats per minute.
* Suffer from asthma, emphysema, bronchitis, kidney disease, pheochromocytoma, diabetes, overactive thyroid, or a history of severe anaphylactic reactions.
* Are scheduled for surgery.

Additionally, participants who meet the inclusion criteria but present with more than one of the following cardiovascular disease (CVD) risk factors will be excluded unless cleared by a cardiologist:

* Family History: Myocardial infarction, coronary revascularization, or sudden death before 55 years of age in a father or male first-degree relative, or before 65 years of age in a mother or female first-degree relative.
* Hypertension: Systolic blood pressure greater than 140 mmHg or diastolic blood pressure greater than 90 mmHg.
* Dyslipidemia: Total serum cholesterol exceeding 200 mg/dl.
* Pre-diabetes: Fasting blood glucose levels between 100 mg/dl and 126 mg/dl.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-24 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Immune Cell Enumeration and Phenotyping | immediately after the intervention
  Whole blood samples will be analyzed for complete blood counts and to quantify lymphocyte and monocyte subtypes using flow cytometry and a comprehensive immunophenotyping panel. This panel is designed to identify major immune cell populations, as well as markers related to differentiation, exhaustion, migration, activation, and inhibition. Specific cell types expressing a surface protein, or combinations of surface proteins, will be reported as the percentage of cells positive for expression and/or by mean fluorescent intensity (MFI). For descriptive purposes, the cell counts of all major lymphocyte and monocyte subtypes will be expressed as cells per microliter (cells/µL) of whole blood. Additionally, isolated peripheral blood mononuclear cells (PBMCs) and expanded cell products will be quantified and phenotyped in a similar manner.
Cytolysis in vitro | immediately after the intervention
  We will assess whether lymphocytes collected during or after exercise, as well as cell products manufactured from these lymphocytes, are more effective at killing hematologic cancer target cells. Using in vitro assays, such as flow cytometry and bioluminescence-based assays, we will compare the cytolytic activity of both the collected lymphocytes and the manufactured cell products to those obtained under resting conditions. Results will be measured as the time required to achieve 10%, 20%, 30%, 40%, and 50% cytolysis, or as the percentage of target cells killed at specific time points (e.g., 4, 8, 24, and 48 hours). We will also evaluate the impact of combination therapies, such as monoclonal antibodies targeting the tumor model, as appropriate.
Tumor Burden and Tumor Free Survival | up to 120-days
  Tumor burden will be evaluated in immunocompromised mice engrafted with human tumors by measuring the size, number, and progression of tumors using imaging techniques such as bioluminescence, MRI, or CT scans, along with physical measurements where applicable. Overall tumor burden will be assessed through metrics like peak tumor size and photon intensity in bioluminescence imaging. Tumor-free survival will be defined as the time from treatment until either the recurrence of detectable tumors or the last follow-up without tumor recurrence. Data will be reported as overall tumor reduction (e.g., percentage decrease in tumor size or number), peak tumor burden, and photon intensity, as well as the duration of tumor-free survival in days. Additional analyses will explore the effects of treatment on delaying tumor progression and improving overall survival.
Clinical xGvHD Score | up to 120-days
  The development of xGvHD (xenogeneic graft-versus-host disease) will be assessed using a clinical scoring system with a possible aggregate score ranging from 0 to 10. Animals will be monitored regularly, and a total score of 5 or higher on two consecutive assessment days will indicate the presence of moderate xGvHD. This scoring system allows for the systematic evaluation of disease severity and progression in response to treatment.
Survival | up to 120 days
  Survival will be monitored as a critical endpoint in this study. Death will be recorded when any of the following criteria are met: (1) the animal experiences greater than 20% weight loss compared to its baseline weight at two consecutive weigh-ins, indicating significant deterioration in health; or (2) the animal exhibits signs of severe morbidity, characterized by an xGvHD score exceeding 7. These criteria ensure that any adverse effects related to treatment or disease progression are accurately captured, allowing for a comprehensive assessment of the survival outcomes in the context of xGvHD.

SECONDARY OUTCOMES:
Single-Cell Secretome | immediately after the intervention
  We will assess the functional phenotype of purified cell types, including CD4+ and CD8+ T cells as well as natural killer (NK) cells, isolated from blood lymphocytes or expanded cell products. This will be accomplished using the Isoplexis single-cell platform and a multiplexed analysis of over 32 cytokines. Polyfunctionality will be evaluated by quantifying the number of distinct cytokines secreted by individual cells (ranging from 0 to 32) after a culture period of 4 to 18 hours. Each assay will include controls: unstimulated cells as a negative control, tumor cells to represent a target, and phorbol myristate acetate (PMA) as a positive control.
CITE-Seq Analysis of Immune Cell Populations | immediately after the intervention
  We will use CITE-Seq to analyze transcriptional and surface protein differences in key human immune cell populations in response to exercise, with and without in vitro tumor challenge. Cell clusters will be annotated using the Azimuth package based on reference human PBMCs. Additionally, we will conduct differential gene expression (DE) analysis and perform Gene Set Enrichment Analysis (GSEA) using Gene Ontology (GO) and Kyoto Encyclopedia of Genes and Genomes (KEGG) terms, applying fold-change and difference metrics for all major immune cell clusters defined by the Azimuth multimodal atlas. We will also sequence various chains of the T-cell receptor (alpha, beta, gamma and delta) to determine T-cell clonal characteristics and antigen specificity using public databases (e.g. VDJdb).
Human Cell Engraftment and Immune Reconstitution: | up to 120-days
  In xenogeneic mice, peripheral blood counts and flow cytometry will be performed on days +7, +14, +21, +28, and +35 following tail bleeding into heparinized capillary tubes. This will assess human CD45+ cell engraftment (% of total human and mouse CD45+ cells) and differences in human immune cell reconstitution using a limited panel of lineage markers due to the restricted blood volumes in mice. If necessary, selected experiments will involve euthanizing mice to evaluate differences in human CD45+ cell and lymphocyte subsets in the bone marrow and spleen.
Pathology and Immunohistochemistry | up to 120-days
  In additional experiments, tissues-including the large and small intestine, liver, lung, and skin-from xenogeneic mice will be harvested for pathological evaluation of xenogeneic graft-versus-host disease (xGvHD). Immunohistochemistry will be performed to assess the types of infiltrating human cells present in the mouse tissues. The quantification of immune cells will be conducted using image analysis software to count the number of positive-staining cells per field of view, allowing for a comparison of immune cell infiltration across different tissues and experimental conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zuniga TM, Baker FL, Smith KA, Batatinha H, Lau B, Gustafson MP, Katsanis E, Simpson RJ. Acute exercise mobilizes NKT-like cells with a cytotoxic transcriptomic profile but does not augment the potency of cytokine-induced killer (CIK) cells. Front Immunol. 2022 Sep 14;13:938106. doi: 10.3389/fimmu.2022.938106. eCollection 2022. PMID 36189306
- [Result] Zuniga TM, Baker FL, Smith KA, Batatinha H, Lau B, Burgess SC, Gustafson MP, Katsanis E, Simpson RJ. Clonal Kinetics and Single-Cell Transcriptional Profiles of T Cells Mobilized to Blood by Acute Exercise. Med Sci Sports Exerc. 2023 Jun 1;55(6):991-1002. doi: 10.1249/MSS.0000000000003130. Epub 2023 Jan 26. PMID 36719647
- [Result] Batatinha H, Diak DM, Niemiro GM, Baker FL, Smith KA, Zuniga TM, Mylabathula PL, Seckeler MD, Lau B, LaVoy EC, Gustafson MP, Katsanis E, Simpson RJ. Human lymphocytes mobilized with exercise have an anti-tumor transcriptomic profile and exert enhanced graft-versus-leukemia effects in xenogeneic mice. Front Immunol. 2023 Apr 3;14:1067369. doi: 10.3389/fimmu.2023.1067369. eCollection 2023. PMID 37077913
- [Result] Baker FL, Smith KA, Mylabathula PL, Zuniga TM, Diak DM, Batatinha H, Niemiro GM, Seckeler MD, Pedlar CR, O'Connor DP, Colombo J, Katsanis E, Simpson RJ. Exercise-induced beta2-adrenergic Receptor Activation Enhances the Antileukemic Activity of Expanded gammadelta T-Cells via DNAM-1 Upregulation and PVR/Nectin-2 Recognition. Cancer Res Commun. 2024 May 13;4(5):1253-1267. doi: 10.1158/2767-9764.CRC-23-0570. PMID 38592213
- [Derived] Batatinha H, Valenzuela AM, Filioglou D, Wilde P, Leite G, Kistner TM, Baker FL, Katsanis E, Simpson RJ. Exercise-Mobilized Lymphocytes Enhance the Function of Cytokine-Induced Memory-like NK-cells Against Myeloid Leukemia. Blood Adv. 2026 Jan 15:bloodadvances.2025018345. doi: 10.1182/bloodadvances.2025018345. Online ahead of print. PMID 41538301